# PERSONALIZING SLEEP INTERVENTIONS TO PREVENT TYPE 2 DIABETES IN COMMUNITY DWELLING ADULTS WITH PREDIABETES: A PHASE 1 SINGLE-CENTER RANDOMIZED CLINICAL TRIAL OF THE EFFECTS OF IMPROVING SLEEP ON GLYCEMIC CONTROL IN PARTICIPANTS WITH PREDIABETES

| ClinicalTrials.gov | 03398902 |
|--------------------|----------|
| Number | 03390902 |

July, 8, 2021

### 1.1 Statistical Hypotheses

Sleep intervention participants will have a lower percentage of time glucose is ≥ 140mg/dL compared to control intervention participants after 8-weeks of treatment.

### 1.2 Analysis Datasets

Primary analyses were performed within an intent-to-treat (ITT) sample, including all participants that were randomized to either the Sleep Intervention or Control Intervention.

# 1.3 Description of Statistical Methods

# 1.3.1 General Approach

The goal of this single site, parallel arm randomized clinical trial was to assess the impact of improved sleep on glycemic control (percent time glucose is ≥ 140) when compared to habitual sleep. Using descriptive analyses, the investigators described each variable using measures of central tendency (means, medians) and variability (standard deviations) for continuous variables; counts and percentages for categorical variables. Data were evaluated for anomalies (e.g., nonrandom missing data, erroneous outliers, multicollinearity, possible confounding) that may invalidate planned analyses.

#### 1.3.2 Analysis of the Primary Efficacy Endpoint(s)

A multivariable Linear regression model was used to assess the effect of the sleep intervention with the subject specific change in the percent time glucose is  $\geq$  140 (Time above target) from baseline as the continuous outcome variable and intervention arm (0=Control Intervention [CI], 1=Sleep Intervention [SI]) as a dichotomous predictor. Effect sizes were presented as beta coefficients and associated 95% confidence intervals, equal to the expected difference between the SI and CI. Important covariates that will be controlled for in these analyses include demographic characteristics including age (continuous), sex (female/male), and race (Asian, Black, White, Other). Statistical significance was determined with a *p*-value < 0.05 using a two-tailed test for significance. Normality was assessed using a skewness cutoff of  $\pm 2$ , following established guidelines.